CLINICAL TRIAL: NCT07068048
Title: Intra-operative Steroid Irrigation for Reducing Recurrent Laryngeal Nerve Palsy Post-thyroidectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Chua Jenna, Master Student, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MREC ID NO: 202456-13711
Record Dates: First submitted 2025-06-23; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Nerve Condition
MeSH Terms: interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-operative Water for Injection for Irrigation for Post-thyroidectomy (Placebo Comparator): For the placebo group, they will received water irrigation over the operative field only which is the current standard of practice at the moment.
  Interventions: Drug: Water for injection
- Intra-operative Dexamethasone Irrigation for Reducing Recurrent Laryngeal Nerve Palsy (Active Comparator): Intra-operatively, all participants recruited must have the recurrent laryngeal nerve identify and confirm with Intraoperative Nerve Monitoring (IONM) device.
  After removal of thyroid gland, 8mg of dexamethasone will be diluted in 100cc of irrigation water and irrigate the operative field for 1 minute for the intervention group.
  Interventions: Drug: Dexametasone

INTERVENTIONS:
Drug: Dexametasone — Intra-operatively, all participants recruited must have the recurrent laryngeal nerve identify and confirm with Intraoperative Nerve Monitoring (IONM) device.
  After removal of thyroid gland, 8mg of dexamethasone will be diluted in 100cc of irrigation water and irrigate the operative field for 1 minute for the intervention group.
  Arms: Intra-operative Dexamethasone Irrigation for Reducing Recurrent Laryngeal Nerve Palsy
Drug: Water for injection — For the placebo group, they will received water irrigation over the operative field only which is the current standard of practice at the moment.
  Arms: Intra-operative Water for Injection for Irrigation for Post-thyroidectomy

SUMMARY:
The main aim of this study is to elucidate whether the topical irrigation of steroid during thyroid surgery can reduce the rate of recurrent laryngeal nerve palsy as majority of nerve dysfunction was due to neuropraxia to axonotmesis.

Intra-operatively, all participants recruited must have the recurrent laryngeal nerve identify and confirm with Intraoperative Nerve Monitoring (IONM) device.

After removal of thyroid gland, 8mg of dexamethasone will be diluted in 100cc of irrigation water and irrigate the operative field for 1 minute for the intervention group.

However for the placebo group, they will received water irrigation over the operative field only which is the current standard of practice at the moment.

Both the otolaryngologist and patient are blinded throughout the whole study.

ELIGIBILITY:
Inclusion Criteria:

* The target population are patients who scheduled for thyroidectomy (include both total or hemithyroidectomy) under UMMC
* Age between 18 years old till 80 years old

Exclusion Criteria:

* Vocal cord paresis before surgery
* No consent
* Allergy towards dexamethasone
* Surgery involved neck dissection
* Retrosternal goitre

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Post thyroidectomy vocal cord assessment will be performed by otolaryngologist within 3 weeks after surgery by using indirect larygoscopy, to look for any vocal cord palsy | Three week post surgery
  if both the vocal cord mobile equally with no phonation gap, indicated no vocal cord palsy if any of the vocal cord paralysed with phonation gap, indicated vocal cord palsy

CONTACTS AND LOCATIONS:
Locations (1):
- UMMC, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT07068048/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT07068048/ICF_001.pdf